CLINICAL TRIAL: NCT06186947
Title: Effects of COVID-19 Infection on Pregnancy Outcomes and Offspring Health: A Large Cohort Study
Brief Title: Effects of COVID-19 Infection on Pregnancy Outcomes and Offspring Health
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Shandong University of Traditional Chinese Medicine (Other); The Second Hospital of Shandong University (Other); The Affiliated Hospital of Qingdao University (Other); Yantai Yuhuangding Hospital Affiliated to Qingdao University (Unknown); Yantai City Yantai Mountain Hospital (Unknown); the First People's Hospital of Jining (Unknown); Weifang People's Hospital (Other); Jining Medical University (Other); Linyi People's Hospital (Other); Dezhou People's Hospital (Other); The Affiliated Hospital of Binzhou Medical College (Unknown); Liaocheng People's Hospital (Other); The Second People's Hospital of Liaocheng (Unknown); Linyi Maternal and Child Healthcare Hospital (Unknown); Heze Hospital of Traditional Chinese Medicine (Unknown); Weihai maternal and child health care hospital (Unknown); Weifang Maternal and Child Health Hospital (Unknown); Tai'an City Central Hospital (Unknown); Zibo Maternal and Child Health Care Hospital (Unknown); Qingdao Women and Children's Hospital (Unknown); The Affiliated Hospital of Shandong University of Traditional Chinese Medicine (Unknown); Qilu Hospital of Shandong University (Other); The Affiliated Hospital of Weifang Medical College (Unknown); Maternal and Child Health Care Hospital of Shandong Province (Unknown); Ren Ji Hospital of Shanghai Jiao Tong University (Unknown)
Responsible Party: Principal Investigator, Chen Zi-Jiang, Academician, Shandong University
Other Study IDs: COVREP
Record Dates: First submitted 2023-12-28; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 group: Patients infected by SARS CoV2 before reproductive events.
  Interventions: Other: No intervention
- Control group: Patients who were not infected by SARS CoV2 before reproductive events.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Participants are not subjected to any specific intervention.

SUMMARY:
This is a large observational cohort study to assess the impact of COVID-19 infection on pregnancy outcomes and offspring health.

DETAILED DESCRIPTION:
The influence of SARS-CoV-2 infection on reproductive outcomes has been uncertain. The goal of this observational study is to assess the impact of COVID-19 infection on pregnancy outcomes and offspring health for patients with childbearing needs.

Participants will:

1. Undergo a questionnaire to gather details on COVID-19 infection history.
2. Provide data about reproductive history.
3. Be invited for physical examination, laboratory tests and ultrasound scans.
4. Undergo a long-term follow up for pregnancy outcome and offspring health.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 18-50 years old.
2. Patients with signed informed consent.
3. Patients with complete COVID-19 infection information.

Exclusion Criteria:

1. Patients with abnormal karyotype
2. Recipients of oocyte donation.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with reproductive needs are recruited for study.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 7 weeks after the day of embryo transfer
  Clinical pregnancy is defined as the ultrasound confirmation of at least one gestational sac.
Ongoing pregnancy rate | 12 weeks after the day of embryo transfer
  Ongoing pregnancy is defined as continued pregnancy beyond 12 weeks of gestation.

SECONDARY OUTCOMES:
Live birth rate | 10 months after the day of embryo transfer
  Live birth is defined as the delivery of any neonate with signs of life at ≥ 28 weeks of gestation.
Pregnancy loss rate | 10 months after the day of embryo transfer
  Pregnancy loss is defined as pregnancy that eventuates in a spontaneous abortion or therapeutic abortion that occurred throughout pregnancy.
Congenital malformation rate | 12 months after the day of embryo transfer
  The number of the malformation neonates/the number of the neonates alive ×100%.

CONTACTS AND LOCATIONS:
Overall Officials: Zi-Jiang Chen, Study Chair — Shandong University
Locations (1):
- Institute of Women, Children and Reproductive Health, Jinan, Shandong, China